CLINICAL TRIAL: NCT04135716
Title: A Prospective, Randomized, Single-blind, Parallel-controlled Multicenter Study Evaluating the Effectiveness of Endo.Angel in Improving the Quality of Colonoscopy
Brief Title: A Multicenter Study Evaluating the Effectiveness of Endo.Angel in Improving the Quality of Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EA-18-003
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Adenoma
MeSH Terms: conditions — Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Randomization results were kept confidential in the general case, and information on the use of EndoAngel was not reflected in the hospital history and documents obtained by other subjects. During the examination and after the examination, researchers should take care to avoid talking to the subjects about random content and avoid unnecessary blindness.
  The evaluator was blinded, and neither the data analysis team nor the pathologist could obtain random result information from the medical history data, regardless of whether the subject used EndoAngel or not.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed group (Experimental): Patients will receive colonoscopy with assistance of Endo.Angel
  Interventions: Diagnostic Test: Colonoscopy with assistance of Endo.Angel
- Non-exposed group (Sham Comparator): Patients will receive colonoscopy without assistance of Endo.Angel
  Interventions: Diagnostic Test: Colonoscopy without assistance of Endo.Angel

INTERVENTIONS:
Diagnostic Test: Colonoscopy with assistance of Endo.Angel — Patients in exposed group will receive colonoscopy with assistance of Endo.Angel,a real-time quality monitoring system based on computer vision,which is used to monitor the velocity of insertion of the endoscope, record the time of insertion and withdrawal of the endoscope, and remind endoscopists of the blind areas caused by intestinal segment slipping.
  Arms: Exposed group
Diagnostic Test: Colonoscopy without assistance of Endo.Angel — Patients in non-exposed group will receive colonoscopy without assistance of Endo.Angel.
  Arms: Non-exposed group

SUMMARY:
Colonoscopy is a key technique in the detection and diagnosis of lower gastrointestinal diseases. High quality endoscopy results in better disease outcomes. However, the operant level of different endoscopists is significantly different.This study aims to construct a real-time quality monitoring system based on computer vision, named Endo.Angel, which is used to monitor the velocity of insertion of the endoscope, record the time of insertion and withdrawal of the endoscope, and remind endoscopists of the blind areas caused by intestinal segment slipping.

DETAILED DESCRIPTION:
This study aims to construct a real-time quality monitoring system based on computer vision, named Endo.Angel, which is used to monitor the velocity of insertion of the endoscope, record the time of insertion and withdrawal of the endoscope, and remind endoscopists of the blind areas caused by intestinal segment slipping.Criteria for inclusion and exclusion are determined prior to endoscopic examination. Candidates who meet all inclusion criteria as well as do not meet all exclusion criteria are bring into the study. Participants randomized before the examination, they are divided into the exposed group assisted by Endo.Angel or the non-exposed group without Endo.Angel. Followup are conducted after the examination.Study will be finished when all followup is done,and the examination result collected from participants will send to an independent review data analysis group.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women over the age of 18 years old;
2. Ability to read, understand and sign informed consent;
3. The investigator believes that the subject understands the flow of the clinical study and is willing and able to complete all the research procedures and follow-up visits in conjunction with the research procedure.

Exclusion Criteria:

1. Colonoscopy patients with absolute contraindications;
2. patients with biopsy contraindications;
3. inflammatory bowel disease, colorectal cancer, history of colorectal surgery;
4. women during pregnancy or lactation;
5. Patients with multiple polyposis syndrome;
6. Patients with known or suspected intestinal obstruction or perforation
7. Previously failed colonoscopy;
8. The investigator believes that the subject is not suitable for high-risk disease or other special conditions in clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1076 (Estimated)
Dates: Start 2019-11-28 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 3 months.
  The numerator is the number of cases of adenoma detected by colonoscopy, and the denominator is the total number of cases of patients undergoing colonoscopy.

SECONDARY OUTCOMES:
The mean number of polyps per procedure | 3 months.
  The numerator is the total number of polyps detected by colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
Polyp Detection Rate | 3 months.
  The numerator is the number of patients with polyps detected by colonoscopy, and the denominator is the total number of patients receiving colonoscopy.
The mean number of adenomas per procedure | 3 months.
  The numerator is the total number of adenomas detected by colonoscopy, and the denominator is the total number of patients undergoing colonoscopy
Detection rate of large, small and minimal polyps | 3 months.
  The numerator was the number of patients with large (≥10 mm), small (4-9 mm), and minimal(≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy
The mean number of large, small and minimal polyps per procedure | 3 months.
  The numerator was the number of large (≥10 mm), small (4-9 mm), and minimal (≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy
Detection rate of large, small and minimal adenomas | 3 months.
  The numerator was the number of patients with large (≥10 mm), small (4-9 mm), and minimal(≤5 mm) adenomas detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China